CLINICAL TRIAL: NCT04522089
Title: A Randomized, Single Center, Open-label, Dose-finding, Phase I Study to Evaluate the Safety and Immunogenicity of Pandemic Virus Vaccine, AdimrSC-2f (SARS-CoV-2), in Healthy Volunteers
Brief Title: A Study to Evaluate the Safety and Immunogenicity of COVID-19 (AdimrSC-2f) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ADPCT20011X
Record Dates: First submitted 2020-08-12; First posted 2020-08-21 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AdimrSC-2f Group 1 (Experimental): low dose mcg
  Interventions: Biological: AdimrSC-2f
- AdimrSC-2f Group 2 (Experimental): low dose mcg+AL
  Interventions: Biological: AdimrSC-2f
- AdimrSC-2f Group 3 (Experimental): medium dose mcg
  Interventions: Biological: AdimrSC-2f
- AdimrSC-2f Group 4 (Experimental): high dose mcg
  Interventions: Biological: AdimrSC-2f

INTERVENTIONS:
Biological: AdimrSC-2f — AdimrSC-2f is a candidate vaccine against COVID-19 developed by Adimmune Corporation (Adimmune). Using the baculovirus-insect cells expression system, the recombinant receptor binding domain (RBD) of SARS-CoV-2 spike (S) protein is amplified and purified. AdimrSC-2f is formulated in the different dosages of Spike (S) protein without/with aluminum content as adjuvant.

SUMMARY:
This study aims to evaluate the safety and immunogenicity of the preventative vaccine, AdimrSC-2f, in healthy volunteers aged from 20 to 60 years old.

DETAILED DESCRIPTION:
The objectives of this phase I study are:

1. to evaluate the safety profile of the AdimrSC-2f vaccine, and
2. to assess the immunogenicity of the AdimrSC-2f vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet ALL inclusion criteria will be included.

  1. Male or non-pregnant female, aged 20 to 60 years old (inclusive).
  2. Subject who is physically and mentally capable of participating the study and are willing to adhere to study procedures.
  3. Subject with no clinically significant abnormal findings in medical history, physical examination, vital signs, or clinical laboratory results at the Screening visit based on the investigator's judgment.
  4. Subject with negative test result in SARS-CoV-2 antibody (IgG and IgM) rapid test at the Screening visit.
  5. Subject with negative serology test results for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, and hepatitis C antibody at the Screening visit.
  6. Subjects' clinical laboratory test results are in the normal range or with abnormal values without clinical significance as judged by the investigator.
  7. Female subject with childbearing potential must have negative result in urine pregnancy test at the Screening visit.
  8. Female subject with childbearing potential must be willing to implement adequate, highly effective contraceptive measure during the study period. Effective birth control includes:

     1. Intrauterine device plus one barrier method
     2. Oral, implantable, or injectable contraceptives plus one barrier method; or
     3. Two barrier methods Effective barrier methods are male or female condoms, diaphragms, or spermicides (creams or gels that contain a chemical to kill sperm). Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for ≥ 1 year.
  9. Male subject who agrees to use an adequate method of contraception during the study period [e.g., barrier contraceptives (male condom)].
  10. Subject who provides informed consent after receiving a detailed explanation of study procedures.

Exclusion Criteria:

* Subjects who meet ANY exclusion criteria will be excluded.

  1. Subject with a body mass index (BMI) < 18.5 kg/m2 (underweight) or ≥ 35 kg/m2 (greater than Class I obesity) at the Screening Visit.
  2. Subject with history of cancer (except localized skin cancer without metastases) within 5 years prior to the Screening visit.
  3. Subject has ongoing or medical history of hypertension or diabetes mellitus.
  4. Subject has ongoing use of tobacco or nicotine-containing products (nicotine patch included) or e-cigarette devices or with history of using nicotine-containing product as documented in medical chart or by verbal confirmation at screening.
  5. Subject with documented history of substance or alcohol abuse in the medical chart or by verbal confirmation within 6 months (approximately 180 days) prior to the Screening visit.
  6. Subject who received any vaccine (live, inactivated, or bacterial) within 1 month (approximately 30 days) prior to the Screening visit.
  7. Subject with hypersensitivity to the ingredients of AdimrSC-2f (including aluminum).
  8. Subject with personal or family history of Guillain-Barré Syndrome.
  9. Subject who has travelled abroad within 3 months (approximately 90 days) prior to the Screening visit.
  10. Subject with influenza-like illness as defined by any of the following symptoms at Screening visit: fever (tympanic temperature ≥ 38℃), dry cough, headache, fatigue, respiratory sputum production (phlegm), dysgeusia, anosmia, shortness of breath, muscle and joint pain, or sore throat.
  11. Female subject who is pregnant or lactating at screening or plans to be pregnant during the study period.
  12. Subject who treated with an investigational drug or device or have participated in a clinical study within 3 months (approximately 90 days) prior to the Screening visit.
  13. Subject with clinically significant abnormal ECG at the Screening visit or with history of clinically significant cardiovascular disease such as arrhythmia, coronary artery disease or heart failure, as judged by the investigator.
  14. Subject with any confirmed or suspected abnormal immune function, immunosuppressive, or immunodeficiency or received any immunosuppressants or immunomodulators within 6 months (approximately 180 days) prior to the Screening visit.
  15. Subject with history of wheezing, asthma, chronic obstructive pulmonary disease, or have used bronchodilator within 3 months (approximately 90 days) prior to the Screening visit.
  16. Subject who had blood donation within 2 weeks prior to the Screening visit.
  17. Subject who received any blood products, including immunoglobulin within 3 months (approximately 90 days) prior to the Screening visit.
  18. Subject who is not suitable to participate in this study as judged by the investigator.
  19. Subject with chronic illness.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
The solicited adverse events (SoAEs) | The 7 days following each vaccination
  Determining the solicited adverse events (SoAEs) (the percentage, severity, and relationship to the AdimrSC-2f vaccine) during 7 days following each vaccination.
Incidence of abnormal laboratory tests results | Day 7 after vaccination
  Determining the clinically significant changes in hematology, biochemistry, and coagulation results from baseline at Visit 2 and Visit 4.

SECONDARY OUTCOMES:
Safety of AdimrSC-2f vaccine: AE | Day 0 to Day 182
  1. Determining the SoAEs and unsolicited AES (the percentage, severity, and relationship to AdimrSC-2f vaccine) during the study period.
  2. Overall AEs and serious adverse events (SAEs) during the study period.
Immunogenicity | Day 7,21,28,and 42
  Determining the changes of antibody titers between baseline and the subsequent scheduled visits
Immunogenicity | Day 21 and 42
  Determining the geometric mean increase (GMI)
Immunogenicity | Day 21 and 42
  Determining the seroconversion rate (SCR)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan